CLINICAL TRIAL: NCT03065218
Title: Evaluation of 99mTc Sestamibi Scans In Patients Who Have Differentiated Thyroid Cancer, Elevated Serum Thyroglobulin Levels, and Negative Diagnostic Imaging Studies
Brief Title: 99mTc Sestamibi Scans In Thyroglobulin Positive Scan Negative Differentiated Thyroid Cancer (DTC) Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-166
Record Dates: First submitted 2016-10-27; First posted 2017-02-27 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Thyroid Cancer
Keywords: Thyroid; sestamibi
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Diseases | interventions — Technetium Tc 99m Sestamibi

STUDY DESIGN:
Intervention Model Description: Clinical evaluation of utility of the FDA approved radiopharmaceutical (i.e., 99mTc sestamibi) for differentiated thyroid cancer in a select patient populaton of patients with elevated serum thyroglobulin levels and negative diagnostic radioiodine scans with the objective of determining utility in identifying the site of metastasis(es) that is accounting for the elevated serum thyroglobulin level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- 99mTc sestamilbi (Experimental): 25 mCi 99mTc sestamibi intravenous injection, once. Then imaged for 45 minutes. More imaging might be required and this will be determined by a nuclear medicine physician onsite
  Interventions: Drug: 99mTc sestamibi

INTERVENTIONS:
Drug: 99mTc sestamibi — The administration of the diagnostic radioisotope, 99mTc sestambi, to image possible metastases in patients with differentiated thyroid cancer.

SUMMARY:
This study is being done to see if the radioisotope 99mTc sestamibi scans can locate what is causing the elevated serum thyroglobulin in persons with differentiated thyroid cancer who have elevated serum thyroglobulin levels and negative diagnostic imaging tests.

This is for patients with:

* Elevated suppressed or stimulated thyroglobulin level (Tg) > 10 ng/ml with or WITHOUT thyroglobulin antibodies ,
* All NEGATIVE standard diagnostic clinical imaging studies (NSDCIS) = negative ultrasound (US), diagnostic radioiodine scan (DRS), chest-x-ray (CXR), computer tomography with or without contrast (CT), and 18F-Fluoro-deoxyglucose positron emission computer tomography scan (18F-FDG PET) within the last 12 mos.
* If EDCIS (extensive diagnostic clinical imaging studies of 18F-sodium fluoride positron emission computer tomography scan (18F NaF PET) or 99mTc methylene diphosphonate bone scan (99mTc MDP), AND negative brain CT or magnetic resonance (MR) are performed, these are also negative.

Voluntary patients will have sestamibi scan performed in 4 phases:

Phase 1: receive an injection into their vein of a radioisotope called 99mTc sestamibi.

Phase 2: wait for 60 to 90 minutes in a waiting room

Phase 3: imaged lying face up on an imaging table while a camera passes around you from the top of the head to approximately the level of knees. This requires approximately 45 minutes

Phase 4: images will be reviewed by the nuclear medicine physician. This will take ~10-15 minutes. If additional images are required to clarify an image, then additional images of that area will be performed on the same camera or an alternate camera. As earlier, the additional images performed lying face up. These images require ~20-45 minutes. The patient will then be released.

The risk of this study is considered very low, and the potential benefits to the patient are considered very high.

DETAILED DESCRIPTION:
This study is being done to see if the radioisotope 99mTc sestamibi scans can locate what is causing the elevated serum thyroglobulin in persons with differentiated thyroid cancer who have elevated serum thyroglobulin levels and negative diagnostic imaging tests.

This is for patients with:

* Elevated suppressed or stimulated thyroglobulin level (Tg) > 10 ng/ml with or WITHOUT thyroglobulin antibodies ,
* All NEGATIVE standard diagnostic clinical imaging studies (NSDCIS), which includes all the following negative studies: ultrasound (US), diagnostic radioiodine scan (DRS), chest-x-ray (CXR), computer tomography with or without contrast (CT), and 18F-Fluoro-deoxyglucose positron emission computer tomography scan (18F-FDG PET) within the last 12 mos.
* If NSDCIS and negative brain CT or magnetic resonance (MR) are performed and are negative, voluntary patients will have 99mTc sestamibi scan performed in 4 phases:

Phase 1: receive an injection into their vein of a radioisotope called 99mTc sestamibi.

Phase 2: wait for 60 to 90 minutes in a waiting room

Phase 3: imaged lying face up on an imaging table while a camera passes around you from the top of the head to approximately the level of knees. This requires approximately 45 minutes

Phase 4: images will be reviewed by the nuclear medicine physician. This will take ~10-15 minutes. If additional images are required to clarify an image, then additional images of that area will be performed on the same camera or an alternate camera. As earlier, the additional images performed lying face up. These images require ~20-45 minutes. The patient will then be released.

Interpretation of 99mTc sestamibi Study.

A. A team of two blinded nuclear medicine physicians will interpret the 99mTc sestamibi, and any area of radioactivity will be graded as by a standard nuclear medicine grading system:

1. Normal physiological activity
2. Probably physiological activity
3. Indeterminate activity
4. Probably metastatic disease
5. Metastatic disease

B. Criteria for "final determination" regarding whether a finding represents physiological activity or metastatic disease:

1. For findings graded as 1 or 2, they will be defined for this study as physiological activity.
2. For findings graded as 3, or 4, the following will be required:

i. Biopsy; however, this will only performed if clinically indicated.

1. Follow-up: It is anticipated that very few biopsies will be performed and because the criteria for entering this study is NDCIS., the only alternative for confirming whether or not a foci of 99mTc sestamibi uptake on a scan is metastases will be follow up, which will be performed on a clinical basis. However, if on follow up any of the following occur, then the focus will be categorized as a metastases (true positive).

1. Subsequent biopsy,
2. Subsequent clinical imaging study(s) (For example, although a lytic bone lesion in the area of interested was not present initially on the CT, a lytic lesion indicative of metastases may subsequently develop in that area, and for this study this will be defined as evidence of metastases of DTC (true positive).

   ii. Blind I-131 treatment** with or without a prefatory scan: If a "blind" I-131 treatment" is clinically selected and the post I-131 therapy scan demonstrates uptake in the same areas as the 99mTc sestamibi, then the finding on the 99mTc sestamibi will be classified for this study as a metastases of DTC.
3. Grade 5 is not anticipated, because unlikely I-131, which can have patterns that are very specific for DTC, 99mTc sestamibi patterns are not specific for DTC.

   * A "blind I-131 treatment" is a potential therapeutic option, and this term means that the treating physician or team cannot identify the source of the patient's elevated Tg, but because of factors such as the level of elevated Tg, the rate of rise of the Tg, and the patient's clinical situation, a therapeutic administration of I-131 is give despite being "blind" to the source of the Tg.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Diagnosed with differentiated thyroid carcinoma;
* At least one prior I-131 therapy, which may be remnant ablation, adjuvant treatment, and/or treatment of distant metastases,
* Elevated suppressed or stimulated thyroglobulin level (Tg) > 10 ng/ml with or WITHOUT thyroglobulin antibodies ,
* All NEGATIVE standard diagnostic clinical imaging studies (SDCIS) = negative ultrasound (US), diagnostic radioiodine scan (DRS), chest-x-ray (CXR), computer tomography with or without contrast (CT), and 18F-Fluoro-deoxyglucose positron emission computer tomography scan (18F-FDG PET) within the last 12 mos.
* If extensive diagnostic clinical imaging studies (EDCIS) of 18F-sodium fluoride positron emission computer tomography scan (18F NaF PET) or 99mTc methylene diphosphonate bone scan (99mTc MDP), AND brain CT or magnetic resonance (MR) are performed, these are also negative.

Exclusion Criteria:

* < 18 years of age;
* Pregnant or breast feeding
* Any SDCIS or EDCIS that is positive and/or suggestive of recurrent and/or distant metastases secondary to DTC. If a study is indeterminate, this will be forwarded to a committee for review and resolution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Van Nostrand, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 99mTc Sestamilbi
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who met study inclusion criteria.
Arm/Group | 99mTc Sestamilbi
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Lesion Detection on 99mTc Sestamibi Study
Description: Any area of radioactivity will be graded by a team of two blinded nuclear medicine physicians to determine if the uptake focus is metastatic disease.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 99mTc Sestamilbi
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: One day after 99mTc Sestamibi administration.
Arm/Group | 99mTc Sestamilbi
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT03065218/Prot_000.pdf
  • Informed Consent Form (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03065218/ICF_001.pdf